CLINICAL TRIAL: NCT04898192
Title: COTEPS: Monitoring of Incidence of Mental Discomfort in the Population of Pregnant Women in the Third Trimester During the Serious COVID-19 Pandemic Conditions
Brief Title: Monitoring of Incidence of Mental Discomfort in Pregnant Women During the Serious COVID-19 Pandemic Conditions
Acronym: COTEPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Comenius University (Other)
Responsible Party: Principal Investigator, Peter Musil, head of project centre Faculty of Medicine, Comenius University
Other Study IDs: EC/045/2021/UNBRuzinov
Record Dates: First submitted 2021-05-21; First posted 2021-05-24 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Pregnant Woman
Keywords: mental state; pregnancy; COVID
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — questionnaire - the complex of 6 questionnaires aimed to recognize the fear of delivery, perinatal anxiety, depressive disorder, obsessive-compulsive disorder, general anxiety disorder, postpartal depression and domestic violence.

SUMMARY:
This study is aimed to detect severe fear of delivery and its association with the incidence of obsessive-compulsive disorder and symptoms of depression and anxiety in the population of pregnant women in the third trimester during the serious COVID-19 pandemic situation in Slovakia. Data will be acquired from three departments of gynaecology and obstetrics of University Hospital Bratislava. The majority of pregnancies from the region are managed in this hospital; the total number of deliveries in 2020 achieved 7,835

DETAILED DESCRIPTION:
The pregnancy is a risk factor for the first manifestation of several mental disorders. Current serious pandemic situation and a constant risk of COVID-19 infection negatively affects the mental state of the population, risk groups of pregnant women in particular. The aim of this project is to discover the incidence of symptoms of depression, anxiety and obsessive-compulsive disorder in association with the fear of delivery in current COVID-19 pandemic conditions in Slovakia. We also decided to add a short tool for detection of domestic violence among other scales to detect the incidence among Slovak pregnant population. All pregnant women in their third trimester who visit the prenatal clinic for their routine weekly check-up will be asked to participate in the study. The questionnaire which comprises of validated mental scales will be handed out to the patients waiting for their examination. After collection of filled questionnaires, those will be later paired with patients' medical documentation and statistically evaluated. The questionnaires will be collected during the period of 1.4.2021-31.3.2022 and statistical analysis will be conducted in the period of 1.4.2022-1.8.2022. It is expected that approximately 1,500 women will be included into the study. All three departments of gynaecology and obstetrics of the University Hospital Bratislava will participate at the study. In total, approximately 7,800 deliveries a year are managed in the University Hospital Bratislava.

Following questionnaires are planned to be used in the study:

* Wijma Delivery Expectancy/Experience Questionnaire - aimed at fear of delivery
* PASS (Perinatal Anxiety Screening Scale) - aimed at anxiety in women before and after delivery
* PHQ-9-SK (Patient Health Questionnaire) - aimed at depressive disorder
* HITS Domestic Violence Screening Tool - aimed at domestic violence
* DOK (The Obsessive-Compulsive Inventory) - aimed at obsessive and compulsive symptoms
* GAD-7 (General Anxiety Disorder-7) - aimed at general anxiety disorder
* EPDS (Edinburgh Postnatal Depression Scale) - aimed at symptoms of postpartal depression

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy after 34th week
* Vital fetus

Exclusion Criteria:

* Unwilling to participate
* Age less than 18 years
* Foetus mortus or perinatal death of the newborn
* Low knowledge of Slovak language
* Serious pathology in the pregnancy (e.g. placenta praevia, known congenital disorders)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant
Study Population: pregnant women in her third trimester who attend regular prenatal check-ups
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
prevalence and risk factors | 9 months
  prevalence and risk factors of depression, anxiety and obsessive-compulsive disorder in the population of pregnant women in association with COVID-19 pandemic situation.

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Zahumensky, prof. MD, Study Chair — Comenius University in Bratislava
Locations (1):
- 2nd Department of Obstetrics and Gynecology, University Hospital Bratislava and Comenius University, Bratislava, Slovak Republic, Bratislava, Slovensko, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided